CLINICAL TRIAL: NCT05505890
Title: Effects of Postoperative Analgesic Modalities on Plasma Creatine Phosphokinase(CPK) Levels After Knee Artroplasty
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SamsunU_SFIPB
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Myotoxicity
Keywords: bupivacaine, myotoxicity, creatine phosphokinase,SFIPB
MeSH Terms: conditions — Myotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SFIPB: suprainguinal fascia iliaca plane block with 50ml of %0.25 bupivacaine will be used for postoperative analgesia
  .
  Interventions: Other: suprainguinal fascia iliaca block
- control: Fascia iliac block will not be applied to this group. Postoperative analgesia will be provided with other analgesia modalities.

INTERVENTIONS:
Other: suprainguinal fascia iliaca block — Suprainguinal fascia iliaca block will be performed after the end of surgery for postoperative analgesia.
  Groups: SFIPB

SUMMARY:
Regional anesthesia and analgesia technics are widely and securely used during orthopedic surgery. Interfascial plane blocks are the latest used ones for analgesia. There are studies in literature indicating that bupivacaine cause myotoxicity. We aimed to examine plasma CPK(creatine phosphokinase) levels to see whether myotoxicity occurs or not after suprainguinal fascial plane block is applied to patients undergoing knee artroplasty surgery.

DETAILED DESCRIPTION:
During 2 months period all elligible patients undergoing knee artoplasty surgery will be included in the study. Different postoperative analgesic modalities will be used according to the anesthesists experience. During routine blood sample tests plasma CPK levels will be tested 3 times of all patients.(preoperative, postoperative 6th hour, postoperative 24th hour) this data will be recorded for 2 months. After this period of time data will be analysed and patients will be grouped according to the analgesic modalities used.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* knee artoplasty patients
* under spinal anesthesia

Exclusion Criteria:

* local anesthetic allergies
* myopathies
* coagulopathies
* Obstructive sleep apne syndrome
* hearth diseases
* liver diseases
* kidney diseases
* thyroid-parathyriod dieseas
* hiperlipidemias using Statins(HMG-CoA reductase inhibitors)
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing knee artroplasty surgery of ASA status 1-3. aged between 18-75years.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
CPK levels | at postoperative 24th hour
  Change from Baseline serum creatine phosphokinase at 24 hours

SECONDARY OUTCOMES:
Number of patients requesting rescue analgesics | up to 24 hours
  Intravenous administration of meperidine 25 mg as a rescue analgesic is planned for patients who complain of severe pain despite multimodal analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Tulgar, Study Chair — Samsun University
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rakhi V, Kaushal S, Singh S. Measurement of bupivacaine induced myotoxicity in interfascial plane blocks: A randomised controlled trial. Indian J Anaesth. 2021 Dec;65(12):886-891. doi: 10.4103/ija.ija_848_21. Epub 2021 Dec 22. PMID 35221361